CLINICAL TRIAL: NCT02688322
Title: Pharmacodynamics Modeling to Optimize Dosage Regimens of Sulbactam in Patients With Acinetobacter Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sutep Jaruratanasirikul (Other)
Collaborators: Prince of Songkla University (Other)
Responsible Party: Sponsor-Investigator, Sutep Jaruratanasirikul, Prince of Songkla Univeersity, Prince of Songkla University
Organization: Prince of Songkla University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SULBAC552011411
Record Dates: First submitted 2016-02-17; First posted 2016-02-23 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2015-01

CONDITIONS: Acinetobacter Infections
Keywords: sulbactam; pharmacokinetics; pharmacodynamics; Acinetobacter infections
MeSH Terms: conditions — Acinetobacter Infections | interventions — Sulbactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 g q12 of sulbactam, 1 h infusion (Experimental): 2 g of sulbactam in 100 ml of normal saline solution was administered via an infusion pump at a constant flow rate 1 h every 12 h.
  Interventions: Drug: Sulbactam

INTERVENTIONS:
Drug: Sulbactam — 2 g in 100 ml of normal saline solution and administered via an infusion pump at a constant flow rate 1 h every 12 h. Blood samples (approximately 5 ml) will be obtained by direct venepuncture at the following time: 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 h after 7th dose of sulbactam

SUMMARY:
Acinetobacter species have emerged as agents of serious nosocomial infections in critically ill patients. Only a few effective antibiotics are currently available for the treatment of this pathogen and, therefore, sulbactam is being considered as an alternative treatment option. The aims of this study were to i) reveal the population pharmacokinetics and ii) assess the probability of target attainment (PTA) of sulbactam in septic critically ill patients caused by Acinetobacter spp. infections.

The study was conducted in septic critically ill patients caused by Acinetobacter spp. Each patient received 2 g every 12 h of sulbactam for 10 days, after which PK studies were carried out on day 4 of sulbactam therapy and a Monte Carlo simulation was performed to determine the probability of attaining a specific pharmacodynamic target.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Patients who had diagnosed an Acinetobacter infections that sensitive to sulbactam and colistin
* Infected at sterile site
* Pneumonia was defined by a new and persistent infiltrate on chest radiography associated with at least one of the following: purulent sputum, temperature>38.3°C or <36°C, a leukocyte count>10,000 cell per mm3, heart rate of >90 beats per min and respiratory rate >20 breaths per min
* Urinary tract infection: Acinetobacter spp ≥ 100,000 cfu/mm3

Exclusion Criteria:

* Patients who are pregnant.
* Patients who have documented hypersensitivity to sulbactam and colistin
* Patients who are chronic renal disease
* Patients who are shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
concentration of sulbactam in plasma | 12 h profile after 7th of sulbactam

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Clinical Pharmacology, Department of Medicine, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand